CLINICAL TRIAL: NCT04487249
Title: A Pilot Randomized Trial Evaluating Short-Term Effectiveness of Vision Therapy in Children With Intermittent Exotropia
Brief Title: Trial of Vision Therapy for Intermittent Exotropia
Acronym: VT-IXT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Stanford University (Other); Ohio State University (Other); Salus University (Other); University of Alabama at Birmingham (Other); Southern College of Optometry (Other); Case Western Reserve University (Other); American Academy of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-08
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Intermittent Exotropia
Keywords: Intermittent Exotropia; Vision Therapy
MeSH Terms: interventions — Orthoptics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vision Therapy (Experimental): Participants will receive 20 consecutive weeks of office-based vision therapy with home therapy.
  Interventions: Other: Vision Therapy
- Observation (No Intervention): Participants will receive no treatment for IXT is received during the study unless one of the deterioration criteria is met.

INTERVENTIONS:
Other: Vision Therapy — 20 consecutive weeks of office-based vision therapy with home therapy that aim to improve the participant's vergence skills, accommodative skills, and sensory fusion.
  Other Names: Orthoptics
  Arms: Vision Therapy

SUMMARY:
The main objective of this randomized trial comparing vision therapy to observation is to determine the short-term effectiveness of vision therapy on distance intermittent exotropia control. The results will help determine whether to proceed to a full-scale, long-term randomized trial.

DETAILED DESCRIPTION:
Vision therapy (VT) is a commonly prescribed treatment for children with intermittent exotropia (IXT). The effectiveness of VT as a treatment modality for children with IXT is unknown because previous studies have largely limited observational or retrospective case series without comparison groups. The objective of this multi-centered pilot randomized trial of VT for IXT compared to observation is to 1) determine the short-term effectiveness of VT on distance intermittent exotropia and 2) determine the feasibility of recruitment and retention of children aged 8 to 16 years old with IXT to participate in a randomized trial of 20 weeks of in-office VT. The results of this trial will provide the needed information to plan and conduct a large-scale randomized trial to determine short-term and long-term effectiveness of VT for IXT in children, with the full-scale randomized trial helping to fill in the gaps in scientific knowledge concerning VT as a treatment for IXT.

ELIGIBILITY:
Major Inclusion Criteria-

* Age 8 - 16 years
* Intermittent exotropia meeting all of the following:

  * Distance exodeviation of 15∆ to 35∆ by prism alternating cover test (PACT)
  * IXT, exophoria, or orthophoria at near
  * Near exodeviation that does not exceed the distance exodeviation by more than 10∆
  * Mean distance control score of 2 points or more with at least one measure being 3 points or higher
  * Mean near control score less than 5 points
* Random dot stereopsis of 200" or better on Preschool Randot Stereotest
* Willingness to accept randomization and no plan to relocate in the next 6 months

Major Exclusion Criteria-

* Treatment for IXT or amblyopia (other than refractive correction) within 3 months prior to enrollment
* Office-based vision therapy for IXT within 6 months prior to enrollment
* Prior office-based vision therapy for IXT of ≥10 sessions
* Prior strabismus, intraocular, or refractive surgery (including BOTOX injection)

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean Distance Control Score | 21 weeks
  The primary analysis will be an intent-to-treat comparison of mean distance control score, determine by the intermittent exotropia office control scale, at outcome using an analysis of covariance model, which will adjust for baseline distance control. The intermittent exotropia office control scale grades the control on a scale of 0 (best control; phoria) to 5 (worst control; constant exotropia).

SECONDARY OUTCOMES:
No Spontaneous Tropia | 21 weeks
  The proportion of participants with no spontaneous tropia at outcome will be compared between treatment groups.No spontaneous tropia is defined as control score of 2 or less on all three assessments of control at distance and near and no exotropia lasting more than 5 seconds throughout the examination.
Change in Distance Control | 21 weeks
  The proportion of participants with >= 1 point change in control and >= 2 points change in control will be compared between treatment groups.

OTHER OUTCOMES:
Change in Vergence and Accommodative Measures | 21 weeks
  The near point of convergence, positive and negative fusional vergence ranges at distance and near, vergence facility, accommodative amplitude, and accommodative facility at outcome will be compared between treatment groups adjusting for the corresponding baseline value. The analysis will be completed separately for each vergence and accommodative measures.
Suppression Status | 21 weeks
  Suppression status will be compared at outcome between treatment groups, adjusting for baseline suppression status. Suppression status when the participant's eyes are in tropic position will be assessed using the suppression scale ranging from 0 (negligible suppression) to 4 (dense suppression).
Objective Eye Movement Recordings | 21 weeks
  Frequency of intermittent exotropia by objective eye movement recordings will be compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Chen, OD, MS, Study Chair — Southern California College of Optometry at Marshall B. Ketchum University
Locations (6):
- United States (6):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - Southern California College of Optometry at Marshall B. Ketchum University, Fullerton, California
  - Stanford University, Stanford, California
  - Ohio State University, Columbus, Ohio
  - Salus University, Philadelphia, Pennsylvania
  - Southern College of Optometry, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No